CLINICAL TRIAL: NCT06325449
Title: Correlating Improvement in PCOS Symptoms to the Percentage of Body Weight Lost in Females Also Living With Obesity - A Prospective Study Using a Multi-disciplinary Multi-modal Approach to Weight-loss
Brief Title: Correlating Improvement in PCOS Symptoms to the Percentage of Body Weight Lost in Females Also Living With Obesity
Acronym: FLOWERS-PCOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: LEAF Weight Loss Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5323
Record Dates: First submitted 2023-11-20; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Polycystic Ovary Syndrome; Obesity
Keywords: Polycystic Ovary Syndrome; Obesity; Endocrine; Noncommunicable Diseases; Surveys and Questionnaires; Metabolic Disease; Insulin Sensitivity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Noncommunicable Diseases; Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Clinic patients with PCOS will be recruited to participate in a 24-week weight loss program. They will all receive the program. There is no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STREAM Weight-loss Program (Experimental): All patients who participate in the study will be recruited to the Intervention Arm and will undergo the STREAM program, a 24-week weight loss program which includes meal replacement, dietician teaching and regular appointments with their bariatric medicine specialist.
  Interventions: Behavioral: STREAM program

INTERVENTIONS:
Behavioral: STREAM program — The STREAM program is a 24-week weight-loss program which includes meal replacement, dietician coaching/teaching and weekly visits with a physician.

SUMMARY:
The goal of this clinical trial is to study the effects of a intensive weight loss program (STREAM) in patients living with PCOS. The main questions the investigators aim to answer are: how much weight will these patients lose over a 24-week program, and what other health markers (ie., insulin sensitivity) will improve and by how much?

Participants will complete a 24-week weight loss program (STREAM). During this program they will:

* weigh themselves
* complete regular bloodwork and
* fill out a Quality of Life questionnaire at regular intervals

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a common disorder affecting up to 20% of women of reproductive age associated with, but not exclusive to, obesity. Excess weight and especially visceral adiposity lead to increased insulin resistance which in turn will promote decreased SHBG concentrations and excess androgen secretion from the ovaries. Weight-loss is known to improve PCOS symptoms in individuals but threshold of weight-loss needed to achieve improvement in many PCOS outcomes is poorly understood, as is the impact of varied weight-loss strategies employed to promote weight loss.

OBJECTIVE The goal of this study is to understand the effects of increasing weight loss thresholds on multiple PCOS symptoms and features, using a 24-week intensive weight loss program (STREAM) with the possibility of added pharmacotherapy for weight loss when indicated.

RESEARCH QUESTION What is the required weight loss to achieve significant improvement in PCOS outcomes including metabolic, endocrine, fertility and mental health parameters? Is there a difference in outcome improvement from different approaches (meal replacement, adjunct pharmacotherapy), independent from weight-loss?

PRIMARY OUTCOMES

To identify the percentage of bodyweight loss needed to achieve significant improvement in each of the following:

* Endocrine parameters (SHBG, Testosterone, Androstenedione, LH/FSH ratio)
* Insulin sensitivity (HOMA-IR)
* Lipid profile (TG, HDL and Non-HDL levels)
* Liver enzyme profile (ALT)
* Menstrual cyclicity (yes/no)
* Quality of life scale (QOLS-public domain, see annex)

STUDY DESIGN Participants will be recruited from those already referred to the LEAF Clinic. Women over the age of 18 who meet the inclusion criteria will be invited to participate in the STREAM program, a 24-week intensive weight-loss program that includes full and partial meal replacement, dietician group coaching and weekly meetings with a weight-loss specialist physician. The program cost, $2250, will be waived for the purpose of limiting sampling bias as the cost can be untenable for many patients.

DATA COLLECTION Participants will complete PCOS-specific blood tests at the launch of the program, at the end of the 24 weeks and then again at 6 months after the program is finished. They will also be asked to complete the same blood draws at every 5% weight loss from their baseline. Participants will also be asked to complete the Quality of Life Scale (QOLS), a short survey, at the same intervals.

ANTICIPATED RESULTS Learning more about individual variations in outcome improvement with gradual weight loss in a population of women living with PCOS will be helpful in individualizing approaches to weight loss in this population. This study could not only help determine predictors of improvement for each outcome but as well identify weight loss strategies that are more efficient for specific outcomes. This will result in better care for women living with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female ≥ 18 years old
* BMI ≥ 30 kg/m2 or ≥ 27 kg/m2 with adiposity-related complications
* English proficiency
* Referral to LEAF Weight Management Clinic

Exclusion Criteria:

* Previous bariatric surgery
* Currently on OCP or using an IUD
* Currently using a pharmacotherapy with an impact on weight (Liraglutide, Semaglutide, Tirzepatide, Naltrexone/Buproprion, Orlistat)
* Currently pregnant
* Currently using an androgen supplement (Testosterone, DHEAS)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Weight will be compared from the beginning of the program, at the end (24 weeks), six months later (52 weeks) and at every major weight loss milestone (5%), a measurement which cannot be done a pre-determined time as weight loss isn't linear/predictable.
  percentage difference in participant weight
Change in Endocrine parameters (EP) as measure by blood test | EP will be compared from the beginning of the program, at the end (24 weeks), six months later (52 weeks) and at every major weight loss milestone (5%), a measurement which cannot be scheduled pre-determined as weight loss isn't predictable.
  Change in blood test results (SHBG, Testosterone, Androstenedione, LH/FSH ratio) which are all endocrine markers of PCOS
Change in insulin sensitivity (IS) as measure by blood test | IS will be compared from the beginning of the program, at the end (24 weeks), six months later (52 weeks) and at every major weight loss milestone (5%), a measurement which cannot be scheduled pre-determined as weight loss isn't predictable.
  Change in blood test results (HOMA-IR) which is a marker of PCOS
Change in Lipid profile (LP) as measure by blood test | LP will be compared from the beginning of the program, at the end (24 weeks), six months later (52 weeks) and at every major weight loss milestone (5%), a measurement which cannot be scheduled pre-determined as weight loss isn't predictable.
  Change in blood test results (TG, HDL and Non-HDL levels) which are markers of PCOS
Change in liver enzyme profile (LEP) as measure by blood test | LEP will be compared from the beginning of the program, at the end (24 weeks), six months later (52 weeks) and at every major weight loss milestone (5%), a measurement which cannot be scheduled pre-determined as weight loss isn't predictable.
  Change in blood test results (ALT) which is a marker of PCOS
Change in Menstrual Cyclicity | Patients will be asked to report on their menstrual cycles at the beginning of the program, at the end (24 weeks), six months later (52 weeks) and at every 5% weightloss milestone, which cannot be scheduled in advance as it isn't predictable/linear.
  Regularity of menstrual cycles
Quality of Life (QoL) Scale | QoLs will be compared from the beginning of the program, at the end (24 weeks), six months later (52 weeks) and at every major weight loss milestone (every 5%) which cannot be done at a predetermined time as weight loss isn't predictable or linear
  QoLs is a public-domain questionnaire measuring several subjective quality-of-life parameters

CONTACTS AND LOCATIONS:
Overall Officials: Judy Shiau, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- LEAF Weight Management Clinic, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers at this time and we are not seeking permission to do so from our research ethics board.